CLINICAL TRIAL: NCT06161584
Title: A Prospective, Multicenter, Open-Label, Observational Phase 4 Study to Evaluate Real-World Safety, Tolerability, and Treatment Patterns of Pegcetacoplan (Syfovre) in Patients With Geographic Atrophy Secondary to Age-Related Macular Degeneration
Status: Active, not recruiting | Type: Observational
Sponsor: Apellis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: APL2-GA-411
Record Dates: First submitted 2023-10-18; First posted 2023-12-08 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-05

CONDITIONS: Geographic Atrophy
MeSH Terms: conditions — Geographic Atrophy | interventions — pegcetacoplan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation
  Interventions: Drug: Pegcetacoplan

INTERVENTIONS:
Drug: Pegcetacoplan — Administered intravitreally (IVT) in eyes with geographic atrophy (GA)
  Other Names: Syfovre

SUMMARY:
A Prospective, Multicenter, Open-Label, Observational Phase 4 Study to Evaluate Real-World Safety, Tolerability, and Treatment Patterns of Pegcetacoplan (Syfovre) in Patients with Geographic Atrophy Secondary to Age-Related Macular Degeneration

ELIGIBILITY:
Inclusion Criteria: Eyes are eligible to be included in the study only if all of the following criteria apply. Ocular-specific inclusion criteria apply to the treated eye(s), unless otherwise specified.

* Eyes that are naive to treatment with pegcetacoplan that are prescribed pegcetacoplan per routine clinical practice according to approved pegcetacoplan prescribing information (ie, the clinical decision to treat with pegcetacoplan must be made before study participation is discussed with the patient)
* Patient age ≥60 years
* Visual acuity better than 20/200 on Snellen chart
* Clinical diagnosis of GA of the macula secondary to AMD in one or both eyes as determined by the investigator using OCT and/or FAF imaging
* GA lesion meeting the following criteria as determined by the investigator's assessment of Spectralis OCT and/or FAF images at screening:

  1. Nonsubfoveal lesion(s)
  2. GA lesion visualized in its entirety on the macula-centered OCT image and not contiguous with any areas of peripapillary atrophy
  3. Presence of any pattern of hyperautofluorescence in the junctional zone of GA; absence of hyperautofluorescence (ie, pattern = none) exclusionary
* Adequate clarity of ocular media and adequate pupillary dilation and fixation to permit the collection of good quality images as determined by the investigator
* Patient willing and able to give informed consent and to comply with the study procedures and assessments

Exclusion Criteria: Ocular-specific exclusion criteria apply to the study eye(s) only, unless otherwise specified.

* GA secondary to a condition other than AMD such as Stargardt disease, cone rod dystrophy, or toxic maculopathies like Plaquenil maculopathy in either eye
* Active, suspected, or history of intraocular inflammation in either eye at screening or on day 1
* Any history of or active choroidal neovascularization associated with AMD or any other cause, including any evidence of retinal pigment epithelial tears or rips in SD OCT imaging
* Presence of an active ocular disease that in the opinion of the investigator compromises or confounds visual function, including but not limited to uveitis and other macular diseases (eg, clinically significant epiretinal membrane, full thickness macular hole, uncontrolled glaucoma/ocular hypertension). Conditions that in the opinion of the investigator are benign, such as peripheral retina dystrophy, are not exclusionary
* Any prior treatment with anti-VEGF agents
* Intraocular surgery (including lens replacement surgery) within 3 months prior to screening
* History of laser therapy in the macular region
* Aphakia or absence of the posterior capsule. Note: Yttrium aluminum garnet laser posterior capsulotomy for posterior capsule opacification done at least 60 days prior to screening is not exclusionary.
* Any ocular condition other than GA secondary to AMD that may require surgery or medical intervention during the study period or, in the opinion of the investigator, could compromise visual function during the study period
* Any contraindication to IVT injection
* Current ocular or periocular infection in either eye
* Intravitreal medical device placement
* Participation in any prior or current systemic experimental treatment within 6 weeks or 5 half lives of the active ingredient (whichever is longer) prior to the start of study treatment or in any other investigational treatments specific to GA. Clinical trials solely involving observation, over-the-counter vitamins, supplements, or diets are not exclusionary
* Medical or psychiatric conditions that, in the opinion of the investigator, make consistent follow-up unlikely or would make the patient an unsafe study candidate
* Known hypersensitivity to fluorescein sodium for injection or hypersensitivity to pegcetacoplan or any of the excipients in pegcetacoplan solution
* History or current use of brolucizumab and/or pharmacological treatments that gain approval for the treatment of GA

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients residing in the United States who are 60 years or older who have geographic atrophy secondary to age-related macular degeneration
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of ocular AEs in treated eyes overall and according to physician-directed treatment interval based on US prescribing information | Up to 36 months
Incidence of other events of interest | Up to 36 months

SECONDARY OUTCOMES:
Assess real-world treatment patterns and use of pegcetacoplan considering the proportion of participants with bilateral GA treated with pegcetacoplan in both eyes | Up to 36 months
If only one eye is treated, the criteria for determination of the eye to be treated | Up to 36 months
The treatment interval (mean days between injections) over time | Up to 36 months
The frequency of imaging on treated eyes (color fundus photography, spectral domain optical coherence tomography [SD-OCT], fundus autofluorescence, optical coherence tomography angiography [OCT-A | Up to 36 months
The treatment adherence to planned dosing frequency: the number of injections administered divided by the number of injections planned | Up to 36 months
The duration of persistence on treatment: continuous medication usage until a gap of ≥3 months | Up to 36 months
The treatment discontinuation and/or switching to other agents approved for treatment of GA | Up to 36 months
The management of new-onset exudative age-related macular degeneration (eAMD) events in eyes treated with pegcetacoplan in clinical practice | Up to 36 months
The proportion of treated eyes that develop eAMD that receive anti-vascular endothelial growth factor (VEGF) injections | Up to 36 months
The number of anti-VEGF injections per month from diagnosis of eAMD | Up to 36 months
The proportion of anti-VEGF injections given on same day in the same eye as pegcetacoplan | Up to 36 months

CONTACTS AND LOCATIONS:
Locations (34):
- United States (34):
  - California Retina Consultants (01-026), Bakersfield, California
  - Retina-Vitreous Associates Medical Group (01-020), Beverly Hills, California
  - Illinois Retina Associates (01-035), Fullerton, California
  - Retinal Consultants Medical Group Inc (01-008), Modesto, California
  - Retina Consultants San Diego Inc. (01-018), Poway, California
  - California Retina Consultants (01-027), Santa Barbara, California
  - Bay Area Retina Associates (01-005), Walnut Creek, California
  - Colorado Retina Associates, PLLC (01-011), Lakewood, Colorado
  - Retina Specialty Institute (01-019), Pensacola, Florida
  - South East Retina Center, PC (01-030), Augusta, Georgia
  - Georgia Retina (01-032), Marietta, Georgia
  - Illinois Retina Associates (01-037), Oak Park, Illinois
  - The Retina Care Center (01-023), Baltimore, Maryland
  - Cumberland Valley Retina Consultants, P.C. (01-002), Hagerstown, Maryland
  - Mid Atlantic Retina Specialist (01-029), Hagerstown, Maryland
  - Retina Consultants of Minnesota, PLLC (01-025), Edina, Minnesota
  - Mid Atlantic Retina Research (01-014), Cherry Hill, New Jersey
  - Mid Atlantic Retina (01-031), Cherry Hill, New Jersey
  - OCLI Research Department (01-007), Oceanside, New York
  - Long Island Vitreoretinal Consultants (01-013), Westbury, New York
  - Western Carolina Retinal Associates, PA (01-009), Asheville, North Carolina
  - Retina Associates of Cleveland, Inc. (01-017), Cleveland, Ohio
  - Retina Associates of Cleveland, Inc. (01-022), Cleveland, Ohio
  - Retina Associates of Cleveland, Inc. (01-016), Youngstown, Ohio
  - Mid Atlantic Retina (01-001), Bethlehem, Pennsylvania
  - The Retina Care Center (01-034) - Satellite Site, York, Pennsylvania
  - Black Hills Regional Eye Institute (01-010), Rapid City, South Dakota
  - Tennessee Retina (01-033), Nashville, Tennessee
  - Integrated Clinical Research (01-024), Abilene, Texas
  - Retina Consultants of Texas (01-004), Bellaire, Texas
  - Texas Retina Associates (01-028), Dallas, Texas
  - Retina Consultants of Texas (01-003), The Woodlands, Texas
  - The Retina Group of Washington (01-021), Fairfax, Virginia
  - Pacific Northwest Retina (01-036), Bellevue, Washington